CLINICAL TRIAL: NCT03266458
Title: Predictive Value of CHA2DS2-VASC Score and Contrast Volume to Creatinine Clearance Ratio in Relation to Mehran Score for Contrast-Induced Nephropathy In ST- Elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ghada morsy, resident at cardiology department at assiut university hospital, Assiut University
Other Study IDs: 17100308
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Contrast-induced Nephropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Primary percutaneous coronary intervention — Urgent percutaneous coronary intervention for ST- elevation myocardial infarction patients.
  Other Names: PPCI

SUMMARY:
all patient presented with ST elevated myocardial infarction and underwent PPCI will be calculated with CHA2DS2-VASC score and contrast volume / creatinine clearance as apredictive value for Contrast induced nephropathy and the predictive value of these scores will be compared with the approved predictive value of MEHRAN score which is also will be calculated to every patient .

DETAILED DESCRIPTION:
Myocardial infarction is a major cause of death and disability worldwide. Coronary reperfusion with primary percutaneous coronary intervention ( PPCI) or fibrinolytic therapy improves outcomes in patients with acute ST elevation myocardial infarction (STEMI).

PPCI can be defined as coronary angioplasty/stenting without prior administration of fibrinolytic agents or GPIIb/IIIa antagonists. These patients are usually treated with aspirin, a loading dose of clopidogrel together with heparin or bivalirudin, before the intervention.

If PPCI is performed promptly, the procedure is superior to fibrinolysis in restoring flow to the infarct-related artery in patients with STEMI.

Current guidelines for the treatment of STEMI recommend a door-to-balloon time of 90 minutes or less for patients undergoing PPCI. Door-to-balloon time has become a performance measure and is the focus of regional and national quality-improvement initiatives.

The contrast induced acute kidney injury has commonly been referred to as contrast induced nephropathy (CIN) defined as an increase in serum creatinine ≥25% or ≥0.5 mg/dl from baseline within 48-72 h after contrast exposure. (Weisbord, et al 2006.

CIN is the third most common cause of hospital-acquired acute kidney injury (AKI) due to impaired renal perfusion and use of nephrotoxic medications.

CIN accounts for 11-12% in all cases of in-hospital AKI, and is also associated with 6% of an overall in-hospital mortality rate.

Severe nephropathy after PCI (caused, at least in part, by radiographic contrast material) occurs in up to 2% of patients.

. It occurs most often among those with cardiogenic shock or underlying renal insufficiency and those of advanced age. . Anaphylactic reactions to radiographic contrast material are very rare. .

Age, left ventricular ejection fraction (LVEF) and estimated glomerular filtration rate (eGFR) are independent predictors of CIN development after PPCI for STEMI. .

CIN is strongly associated with late renal and cardiovascular adverse events. However, excluding peri-procedural hydration and the use of small amounts of low-osmolarity contrast media, few agents have proven to be effective for CIN. .

The identification of high-risk patients and preventive optimal hydration are key measures to reduce the incidence of CIN.

Several studies have assessed the role of contrast volume to creatinie clearance ratio (V/CrCl) as a reliable predictor of CIN with conflicting results and proposing different cut-off values. .

V/CrCl ≥ 6.15 was considered as the best discriminant value for the prediction of CIN, which occurred in 25.1% of patients with V/CrCl ≥ 6.15 versus 9.7% in patients with V/CrCl < 6.15. These results were also confirmed at multivariate analysis after correction for all baseline confounders.

The CHA2DS2-VASC score includes the following variables: congestive heart failure (CHF), hypertension, age ≥75 years, diabetes mellitus (DM), previous stroke, vascular disease, age 65 to 74 years, sex. The score is traditionally used for embolic risk stratification in atrial fibrillation (AF) patients.

The CHA2DS2-VASC score, used for embolic risk stratification in AF, has been reported recently to predict adverse clinical outcomes in patients with acute coronary syndrome (ACS), regardless of having AF.

Kurtul et al.(2016) investigated the correlation between the CHA2DS2-VASC score and CIN in ACS patients who underwent urgent PCI and concluded that CHA2DS2-VASC score can be used as a new, simple and reliable tool to predict CIN in patients with ACS who underwent urgent PCI.

Mehran score is a risk score for the prediction of CIN after PCI and it was reported by Mehran et al. In (2004).

The Mehran score has been the most widely used risk score for predicting the risk of CIN. In recent years, there was a proliferation of new scores and methods to predict CIN (Gao, et al.2014), however, their usefulness and extension to clinical practice is limited. The Mehran CIN score was designed in 2004 and based on its simplicity and because it allows early and correct identification of those individuals at high risk for CIN, it is currently the most widely used tool for predicting the risk of CIN.

That risk score includes 8 prognostic variables: hypotension, use of intra-aortic balloon pump, CHF, age, anaemia, DM, contrast media volume and eGFR.

The aim of the study:

1- To evaluate the role of the contrast volume to creatinine clearance ratio (V/CrCl) and the role of CHA2DS2-VASC score in the prediction of contrast-induced nephropathy after PPCI.

2. To compare the CHA2DS2-VASC score with Mehran risk score for predicting the risk of CIN after PPCI.

3. To detect the best cut-off point of CV/CrCl ratio in our population. Patients and methods

1-Study population: The study will include > 210 patients ( calculated sample size) who have STEMI and undergoing PPCI in Cath lab of Orman university Heart Hospital of Assiut University during the period between January 2018 and December 2018.

The sample size was calculated using Epi-info version 7. Based on previous studies, the incidence of CIN in patients undergoing PPCI for STEMI was 5.2% with a power of 80 and confidence level 95%, worst expected value 2.2%, the sample needed for the study was estimated to be about 210 patient [13].

3- Inclusion and Exclusion criteria

Inclusion criteria:

- All patients with STEMI who are eligible for primary PCI will be enrolled in the study.

Exclusion criteria:

1. If the coronary anatomy was not suitable for PCI.
2. If emergency bypass grafting was required.
3. Patients in chronic peritoneal or hemodialytic treatment. 4- Methods:

All patients will be subjected to:

A. Full history taking: including age, sex, history of DM, HTN, Smoking, dyslipidemia, history of cerebrovascular stroke, family history of renal troubles. Also to assess the onset of chest pain and time to reperfusion.

B. Thorough physical examination:

* General examination including intra-procedural blood pressure and heart rate assessment.
* Chest examination: to define Killip score.
* Cardiac examination to detect signs of heart failure. C. Twelve lead ECG: To diagnose STEMI and follow up. D. Collecting baseline venous blood samples for Random blood glucose, CBC, serum creatinin, GFR, electrolytes and lipogram before the procedure.

E. Coronary angiography and primary PCI will be done by an interventional cardiologist (member of PPCI team). After the procedure TIMI flow of the culprit vessel will be reported, as well as the volume of used contrast material and time of X-ray exposure.

F. Creatinine clearance will be calculated using Cockcroft-Gault formula and calculating CV/CrCl ratio.

G. Echocardiography : will be performed immediately after transfer of the patient to CCU to assess the ejection fraction of the heart ( on admission and before discharge).

H. Daily follow up of serum creatinine at 24, 48 hours. I. CHA2DS2-VASC score will be calculated for each patient. Based on the CHA2DS2-VASC score, patients are given 1 point for CHF, hypertension, age 65 to 74 years, diabetes mellitus, vascular disease and female gender and 2 points for age 75 years or older and previous stroke or transient ischemic attack.

I. Mehran risk score will be calculated, that risk score includes 8 prognostic variables: hypotension (5 points, if systolic blood pressure <80 mmHg for at least 1 hour requiring inotropic support), use of intra-aortic balloon pump (5 points), CHF (5 points, if class III/IV by New York Heart Association Classification or history of pulmonary edema), age (4 points, if >75 years), anemia (3 points, if hematocrit <39% for men and <36 for women), diabetes mellitus (3 points ), contrast media volume (1 point per 100 ml), and estimated GFR 2 points, if GFR 60 to 40 ml/min per 1.73 m2; 4 points, if GFR 40 to 20; 6 points, if GFR <20).

Four categories of CIN risk of were established from the cut-off points and intervals defined by Mehran et al. 2010 as follow:

1. Low, <5 points.
2. Moderate, 6 to 10 points.
3. High, 11 to 15 points.
4. Very high, >15 points.
5. Statistical analysis:

Statistical analysis will be performed using the SPSS 20.0 statistical package. All enrolled patients will be divided into two groups according to CHA2DS2-VASC score. Clinical, laboratory, and procedural data will be compared with the use of Student t or Mann-Whitney U test for continuous variables (expressed as mean ± standard deviation for parametric variables, and median and interquartile ranges [25-75 percentile levels] for nonparametric variables) and chi-square test for categorical variables ( expressed as counts and percentages).

Receiver operating characteristic (ROC) curves will be used to identify the optimum cut-off values of V/CrCl ratio and CHA2DS2-VASC score and the number of CHA2DS2-VASC score to predict the development of CIN.

Multiple logistic regression analysis will be performed to evaluate the relationship between the Faculty of Medicine Institutional Review Board (IRB) Assiut Medical School Research Proposal Form 11 V/CrCl value or CHA2DS2-VASC score and the incidence of CIN, after correction for baseline confounding factors (clinical and demographic variables with a P-value<0.05), which will be entered in the model in block .

ELIGIBILITY:
Inclusion Criteria:

* All patients with STEMI who are eligible for primary PCI will be enrolled in the study.

Exclusion Criteria:

* (1) If the coronary anatomy was not suitable for PCI. (2) If emergency bypass grafting was required. (3) Patients in chronic peritoneal or hemodialytic treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include > 210 patients ( calculated sample size) who have STEMI and undergoing PPCI in Cath lab of Orman university Heart Hospital of Assiut University starting from January 2018 .
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Contrast induced nephropathy | 48 hours
  contrast induced nephropathy (CIN) defined as an increase in serum creatinine ≥25% or ≥0.5 mg/dl from baseline within 48 h after contrast exposure so we will follow up creatinine level according to the defenition .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Mehran R, Brar S, Dangas G. Contrast-induced acute kidney injury. Underappreciated or a new marker of cardiovascular mortality? J Am Coll Cardiol. 2010 May 18;55(20):2210-1. doi: 10.1016/j.jacc.2009.12.051. No abstract available. PMID 20466201
- [Background] Amin AP, Salisbury AC, McCullough PA, Gosch K, Spertus JA, Venkitachalam L, Stolker JM, Parikh CR, Masoudi FA, Jones PG, Kosiborod M. Trends in the incidence of acute kidney injury in patients hospitalized with acute myocardial infarction. Arch Intern Med. 2012 Feb 13;172(3):246-53. doi: 10.1001/archinternmed.2011.1202. PMID 22332157
- [Background] Ando G, Morabito G, de Gregorio C, Trio O, Saporito F, Oreto G. Age, glomerular filtration rate, ejection fraction, and the AGEF score predict contrast-induced nephropathy in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention. Catheter Cardiovasc Interv. 2013 Nov 15;82(6):878-85. doi: 10.1002/ccd.25023. Epub 2013 Jun 27. PMID 23703775
- [Background] Ando G, Morabito G, de Gregorio C, Trio O, Saporito F, Oreto G. The ACEF score as predictor of acute kidney injury in patients undergoing primary percutaneous coronary intervention. Int J Cardiol. 2013 Oct 9;168(4):4386-7. doi: 10.1016/j.ijcard.2013.05.049. Epub 2013 May 24. No abstract available. PMID 23711447
- [Background] Anthopoulos, P., I. Antonellis, et al. (2009).
- [Background] Bartholomew BA, Harjai KJ, Dukkipati S, Boura JA, Yerkey MW, Glazier S, Grines CL, O'Neill WW. Impact of nephropathy after percutaneous coronary intervention and a method for risk stratification. Am J Cardiol. 2004 Jun 15;93(12):1515-9. doi: 10.1016/j.amjcard.2004.03.008. PMID 15194023
- [Background] Bartorelli AL, Marenzi G. Contrast-induced nephropathy. J Interv Cardiol. 2008 Feb;21(1):74-85. doi: 10.1111/j.1540-8183.2007.00318.x. Epub 2007 Dec 12. PMID 18086132
- [Background] Barbieri L, Verdoia M, Marino P, Suryapranata H, De Luca G; Novara Atherosclerosis Study Group. Contrast volume to creatinine clearance ratio for the prediction of contrast-induced nephropathy in patients undergoing coronary angiography or percutaneous intervention. Eur J Prev Cardiol. 2016 Jun;23(9):931-7. doi: 10.1177/2047487315614493. Epub 2015 Nov 2. PMID 26525064
- [Background] Cho JY, Jeong MH, Hwan Park S, Kim IS, Park KH, Sim DS, Yoon NS, Yoon HJ, Park HW, Hong YJ, Kim JH, Ahn Y, Cho JG, Park JC, Kang JC. Effect of contrast-induced nephropathy on cardiac outcomes after use of nonionic isosmolar contrast media during coronary procedure. J Cardiol. 2010 Nov;56(3):300-6. doi: 10.1016/j.jjcc.2010.07.002. Epub 2010 Aug 13. PMID 20708903
- [Background] Fox CS, Muntner P, Chen AY, Alexander KP, Roe MT, Wiviott SD. Short-term outcomes of acute myocardial infarction in patients with acute kidney injury: a report from the national cardiovascular data registry. Circulation. 2012 Jan 24;125(3):497-504. doi: 10.1161/CIRCULATIONAHA.111.039909. Epub 2011 Dec 16. PMID 22179533
- [Background] Furman MI, Dauerman HL, Goldberg RJ, Yarzebski J, Lessard D, Gore JM. Twenty-two year (1975 to 1997) trends in the incidence, in-hospital and long-term case fatality rates from initial Q-wave and non-Q-wave myocardial infarction: a multi-hospital, community-wide perspective. J Am Coll Cardiol. 2001 May;37(6):1571-80. doi: 10.1016/s0735-1097(01)01203-7. PMID 11345367
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Keeley EC, Hillis LD. Primary PCI for myocardial infarction with ST-segment elevation. N Engl J Med. 2007 Jan 4;356(1):47-54. doi: 10.1056/NEJMct063503. No abstract available. PMID 17202455
- [Background] Kelly AM, Dwamena B, Cronin P, Bernstein SJ, Carlos RC. Meta-analysis: effectiveness of drugs for preventing contrast-induced nephropathy. Ann Intern Med. 2008 Feb 19;148(4):284-94. doi: 10.7326/0003-4819-148-4-200802190-00007. PMID 18283206
- [Background] Le May MR, So DY, Dionne R, Glover CA, Froeschl MP, Wells GA, Davies RF, Sherrard HL, Maloney J, Marquis JF, O'Brien ER, Trickett J, Poirier P, Ryan SC, Ha A, Joseph PG, Labinaz M. A citywide protocol for primary PCI in ST-segment elevation myocardial infarction. N Engl J Med. 2008 Jan 17;358(3):231-40. doi: 10.1056/NEJMoa073102. PMID 18199862
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] Mahmoud, K. S., Ibrahem, A. M., Saad, M., & Awny, M. (2014). Relation between serum B-type brain natriuretic peptide level and complexity & severity of coronary artery disease in non-ST elevation myocardial infarction. The Egyptian Heart Journal, 66(3), 263-268.
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Mehta RH, Harjai KJ, Grines L, Stone GW, Boura J, Cox D, O'Neill W, Grines CL; Primary Angioplasty in Myocardial Infarction (PAMI) Investigators. Sustained ventricular tachycardia or fibrillation in the cardiac catheterization laboratory among patients receiving primary percutaneous coronary intervention: incidence, predictors, and outcomes. J Am Coll Cardiol. 2004 May 19;43(10):1765-72. doi: 10.1016/j.jacc.2003.09.072. PMID 15145097
- [Background] Menees DS, Peterson ED, Wang Y, Curtis JP, Messenger JC, Rumsfeld JS, Gurm HS. Door-to-balloon time and mortality among patients undergoing primary PCI. N Engl J Med. 2013 Sep 5;369(10):901-9. doi: 10.1056/NEJMoa1208200. PMID 24004117
- [Background] Nikolsky E, Aymong ED, Halkin A, Grines CL, Cox DA, Garcia E, Mehran R, Tcheng JE, Griffin JJ, Guagliumi G, Stuckey T, Turco M, Cohen DA, Negoita M, Lansky AJ, Stone GW. Impact of anemia in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention: analysis from the Controlled Abciximab and Device Investigation to Lower Late Angioplasty Complications (CADILLAC) Trial. J Am Coll Cardiol. 2004 Aug 4;44(3):547-53. doi: 10.1016/j.jacc.2004.03.080. PMID 15358018
- [Background] Piper WD, Malenka DJ, Ryan TJ Jr, Shubrooks SJ Jr, O'Connor GT, Robb JF, Farrell KL, Corliss MS, Hearne MJ, Kellett MA Jr, Watkins MW, Bradley WA, Hettleman BD, Silver TM, McGrath PD, O'Mears JR, Wennberg DE; Northern New England Cardiovascular Disease Study Group. Predicting vascular complications in percutaneous coronary interventions. Am Heart J. 2003 Jun;145(6):1022-9. doi: 10.1016/S0002-8703(03)00079-6. PMID 12796758
- [Background] Sadeghi HM, Stone GW, Grines CL, Mehran R, Dixon SR, Lansky AJ, Fahy M, Cox DA, Garcia E, Tcheng JE, Griffin JJ, Stuckey TD, Turco M, Carroll JD. Impact of renal insufficiency in patients undergoing primary angioplasty for acute myocardial infarction. Circulation. 2003 Dec 2;108(22):2769-75. doi: 10.1161/01.CIR.0000103623.63687.21. Epub 2003 Nov 24. PMID 14638545
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Shusterman N, Strom BL, Murray TG, Morrison G, West SL, Maislin G. Risk factors and outcome of hospital-acquired acute renal failure. Clinical epidemiologic study. Am J Med. 1987 Jul;83(1):65-71. doi: 10.1016/0002-9343(87)90498-0. PMID 3605183
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. J Am Coll Cardiol. 2007 Nov 27;50(22):2173-95. doi: 10.1016/j.jacc.2007.09.011. No abstract available. PMID 18036459
- [Background] Tofield A. Pharmaco-invasive vs. facilitated percutaneous coronary intervention strategies for ST-segment-elevation acute myocardial infarction patients in the new ESC Guidelines. Eur Heart J. 2009 Dec;30(23):2817. doi: 10.1093/eurheartj/ehp409. No abstract available. PMID 19952008
- [Background] Weisbord SD, Chen H, Stone RA, Kip KE, Fine MJ, Saul MI, Palevsky PM. Associations of increases in serum creatinine with mortality and length of hospital stay after coronary angiography. J Am Soc Nephrol. 2006 Oct;17(10):2871-7. doi: 10.1681/ASN.2006030301. Epub 2006 Aug 23. PMID 16928802
- [Background] Wi J, Ko YG, Kim JS, Kim BK, Choi D, Ha JW, Hong MK, Jang Y. Impact of contrast-induced acute kidney injury with transient or persistent renal dysfunction on long-term outcomes of patients with acute myocardial infarction undergoing percutaneous coronary intervention. Heart. 2011 Nov;97(21):1753-7. doi: 10.1136/hrt.2010.218677. Epub 2011 May 20. PMID 21602521
- [Background] Zheng ZJ, Croft JB, Giles WH, Mensah GA. Sudden cardiac death in the United States, 1989 to 1998. Circulation. 2001 Oct 30;104(18):2158-63. doi: 10.1161/hc4301.098254. PMID 11684624
- [Background] Kurtul A, Yarlioglues M, Duran M. Predictive Value of CHA2DS2-VASC Score for Contrast-Induced Nephropathy After Percutaneous Coronary Intervention for Acute Coronary Syndrome. Am J Cardiol. 2017 Mar 15;119(6):819-825. doi: 10.1016/j.amjcard.2016.11.033. Epub 2016 Dec 18. PMID 28040187
- [Background] Chen SL, Zhang J, Yei F, Zhu Z, Liu Z, Lin S, Chu J, Yan J, Zhang R, Kwan TW. Clinical outcomes of contrast-induced nephropathy in patients undergoing percutaneous coronary intervention: a prospective, multicenter, randomized study to analyze the effect of hydration and acetylcysteine. Int J Cardiol. 2008 Jun 6;126(3):407-13. doi: 10.1016/j.ijcard.2007.05.004. Epub 2007 Jul 24. PMID 17651830